CLINICAL TRIAL: NCT00448604
Title: Impact of Viral Infections in Patients With Chronic Obstructive Pulmonary Diseases: Virological Work-up During Exacerbations and 1-year Follow-up
Brief Title: Viral Infections in Chronic Obstructive Pulmonary Disease (COPD) Exacerbations
Acronym: VICE
Status: Completed | Type: Observational
Sponsor: University Hospital, Geneva (Other)
Collaborators: Ligue Pulmonaire Genevoise (Other)
Responsible Party: O. Rutschmann, HUG, Geneva
Other Study IDs: 06-257
Record Dates: First submitted 2007-03-16; First posted 2007-03-19 (Estimated); Last update posted 2010-11-04 (Estimated); Status verified 2009-02

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Respiratory Tract Infections; Virus Diseases; Lung Diseases, Obstructive
Keywords: procalcitonin; acute exacerbation; RT-PCR; Biological Markers
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Respiratory Tract Infections; Virus Diseases; Lung Diseases, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Naso-pharyngeal swaps
Oversight: Data Monitoring Committee: No

SUMMARY:
The objectives of the study are

* to determine the prevalence of respiratory virus infections in COPD patients, during and outside acute exacerbation
* to explore the impact of these viral infections on the outcome of these patients
* to explore the association between blood procalcitonin levels and viral infections in this population.

DETAILED DESCRIPTION:
Background

Chronic obstructive pulmonary disease (COPD) is a leading cause of morbidity due to repeated exacerbations. The impact of viral infections during and outside COPD exacerbations is poorly understood and there is only scarce data on the role of new biological markers of infection for the management of COPD exacerbations.

Objectives of the project

The investigators aim to

1. describe the epidemiology of viral infections in patients admitted with an exacerbation of their COPD;
2. explore the evolution of viral infections outside exacerbations;
3. analyze the impact of viral infections on clinical outcomes;
4. explore the role of biological markers (CRP, procalcitonin) for the diagnosis and prognosis of viral infections.

Methods

The investigators will prospectively follow-up 100 patients admitted with an acute exacerbation of their COPD. Virological samples will be obtained at admission and at 3 months, to explore the evolution outside episodes of acute exacerbation. Clinical information will be obtained after one-year follow-up. Samples will be tested by RT-PCR for 15 respiratory viruses. The impact of viral infections and the role of biological markers will be explored using univariate and multivariate Cox proportional hazard models.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive patients known or suspected for moderate to very severe COPD and admitted in the emergency center for an acute exacerbation of their COPD
* Age above 18 years
* We plan to include 100 patients with a complete work-up and follow-up
* Written informed consent will be obtained from every participant

Exclusion Criteria:

* Patients requiring oro-tracheal intubation
* Patients unable to give their informed consent due to their clinical condition
* Other obvious cause of dyspnea (pulmonary embolism, acute pulmonary edema, lobar pneumonia)
* Patients suffering from bronchiectasis, asthma, pulmonary fibrosis and mineral dust pneumoconiosis
* Patients with a history of active tuberculosis
* Patients with a history of ischemic cerebral stroke and subsequent deglutition dysfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with COPD admitted with acute exacerbation
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2007-05; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Olivier T Rutschmann, MD, MPH, Principal Investigator — University Hospital, Geneva
Locations (1):
- Geneva University Hospital, Geneva, Canton of Geneva, Switzerland

REFERENCES:
- [Derived] Kherad O, Kaiser L, Bridevaux PO, Sarasin F, Thomas Y, Janssens JP, Rutschmann OT. Upper-respiratory viral infection, biomarkers, and COPD exacerbations. Chest. 2010 Oct;138(4):896-904. doi: 10.1378/chest.09-2225. Epub 2010 Apr 30. PMID 20435659